CLINICAL TRIAL: NCT03625960
Title: Trichloroacetic Acid Versus Cantharone for the Treatment of Perenial Warts
Brief Title: Cantharone for the Treatment of Perenial Warts
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: University of California, San Francisco (Other); St Vincent's Hospital (Other)
Responsible Party: Principal Investigator, Maurice-Andre Recanati, Assistant Professor, Clinical Educator, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01551
Record Dates: First submitted 2018-08-02; First posted 2018-08-10 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Wart, Genital
Keywords: warts; trichloroacetic acid
MeSH Terms: conditions — Condylomata Acuminata; Warts | interventions — Cantharidin; Trichloroacetic Acid

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to receive either trichloroacetic acid or cantharidine treatment.
Who Masked: Investigator
Masking Description: Patients will be randomized to receive treatment with trichloroacetic acid or cantharidine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cantharidine group (Experimental): Application of cantharidine to perenial warts
  Interventions: Drug: Cantharidin
- trichloroacetic acid group (Active Comparator): application of trichloroacetic acid to perenial warts
  Interventions: Drug: Trichloroacetic Acid

INTERVENTIONS:
Drug: Cantharidin — A thin film of cantharidin is applied to the surface of the wart and to 1 millimeter area surrounding the wart. After the film dries, it is covered with an occlusive dressing for 24 hours. The patient removes the area the next day and thoroughly washes the area with soap and water. Patients return to clinic a week later.
  Arms: Cantharidine group
Drug: Trichloroacetic Acid — Trichloroacetic acid is applied to the surface of the wart with a wooden applicator and after drying the area is washed with soap and water in an hour.
  Arms: trichloroacetic acid group

SUMMARY:
Comparison of trichloroacetic acid versus cantharidine for the treatment of perenial warts.

DETAILED DESCRIPTION:
Warts are one of the most common sexually transmitted diseases. They are caused by the human papilloma virus (HPV) that causes cervical cancer. Warts can grow, obstruct labor, and spread. Patients presenting to the obgyn clinic with perenial warts were randomized to treatment with trichloroacetic acid (one of the many types of treatments) or to the treatment with cantharidine group. Cantharidine is a vesicant extracted from beetle bugs which painlessly causes a small blister to form and cures the patient from the HPV infection causing the wart . We compared cosmesis, scar formation, pain and number of treatments (visits) as well as effectiveness in both groups.

Objectives

1. Determine if cantharone is more effective than trichloroacetic acid (TCA) for removal of warts
2. Compare pain levels (pain during application) for each method
3. Compare patient satisfaction for each method
4. Compare scar formation and cosmesis for each method

ELIGIBILITY:
Inclusion Criteria:

* Warts on the perenial area
* Less than 4mm across.

Exclusion Criteria:

* Pregnancy
* Less than 18 years old
* Lesions larger than 4 millimeters across
* Unclear diagnosis
* Internal warts
* Diabetes
* HIV
* Warts within 2 cm of mucosal areas

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — This is a study on perenial genital warts, near the vulvovaginal area. Only women have vulvovaginas.
Enrollment: 12 (Actual)
Dates: Start 2006-06-15 (Actual); Primary Completion 2007-06-15 (Actual); Study Completion 2007-07-15 (Actual)

PRIMARY OUTCOMES:
Pain on treatment | at 30 minutes time point from application of treatment.
  Comparison of pain when treatment is applied. The patient is asked on a scale of 0-5 (with 5 being extreme pain, 4 being severe pain, 3 being moderate, 2 being mild, 1 being slight and zero being no pain, how do you rate your pain.

SECONDARY OUTCOMES:
Assessment of a patient's likelihood of using this method again as measured on a survey question | 2 weeks from starting therapy
  A questionnaire given to the patient at the conclusion of the study and containing the question "on a scale from 1-5 (5 most likely) how likely are you to recommend this method to a friend or using it again yourself".
Presence of scarring or skin discoloration | 2 weeks from starting therapy
  At the time of wart eradication, the treatment area is examined for healing. The clinician rates cosmesis on a scale from 0-5 with 5-skin grows back perfectly, 4-slight discoloration, 3-thickened skin, 1-slight scarring and 0-scarring.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bakardzhiev I, Kovachev E. [Comparative assessment of the methods of treatment of Condylomata acuminata]. Akush Ginekol (Sofiia). 2011;50(4):45-51. Bulgarian. PMID 22479897
- [Result] Kollipara R, Ekhlassi E, Downing C, Guidry J, Lee M, Tyring SK. Advancements in Pharmacotherapy for Noncancerous Manifestations of HPV. J Clin Med. 2015 Apr 24;4(5):832-46. doi: 10.3390/jcm4050832. PMID 26239450
- [Result] EPSTEIN WL, KLIGMAN AM. Treatment of warts with cantharidin. AMA Arch Derm. 1958 May;77(5):508-11. doi: 10.1001/archderm.1958.01560050014003. No abstract available. PMID 13519856
- [Result] Ramirez-Fort MK, Au SC, Javed SA, Loo DS. Management of cutaneous human papillomavirus infection: pharmacotherapies. Curr Probl Dermatol. 2014;45:175-85. doi: 10.1159/000356069. Epub 2014 Mar 13. PMID 24643186